CLINICAL TRIAL: NCT00600041
Title: Heart Issues of PantoPrazOle (HIPPO)
Brief Title: Placebo-Controlled Crossover Study for the Investigation of the Effect of Pantoprazole on Cardiac Contractility
Acronym: HIPPO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Herzzentrum Goettingen (Other)
Collaborators: University of Göttingen (Other); Gastroenterology and Endocrinology, University Medicine of Goettingen (Other); Medical Statistics, University Medicine of Goettingen (Other)
Responsible Party: Gerd Hasenfuss/Prof. Dr., Head of dept. of Cardiology and Pneumology, Herzzentrum Goettingen, Dept. of Cardiology and Pneumology
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HIPPO1-2004-11-01; 2004-004355-18 (EudraCT)
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Last update posted 2009-03-24 (Estimated); Status verified 2008-02

CONDITIONS: Healthy
Keywords: Proton Pump Inhibitors; pantoprazole; Cardiac Output; Echocardiography; adverse effects
MeSH Terms: interventions — Pantoprazole; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Pantoprazole IV
  Interventions: Drug: Pantoprazole
- B (Placebo Comparator): NaCl 0.9% IV
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pantoprazole — 80 mg IV over 2 minutes, followed by 8 mg/h IV for 60 minutes
  Other Names: Pantozol i.v.; Protonix I.V.
  Arms: A
Drug: Placebo — Identical infusion manner like experimental arm
  Other Names: NaCl 0.9%
  Arms: B

SUMMARY:
Recently, negative inotropy of pantoprazole has been shown in isolated human myocardium. This study was designed to test the clinical relevance of this finding in healthy volunteers by measuring left ventricular function during infusion of a common intravenous high dose regimen of pantoprazole.

DETAILED DESCRIPTION:
Purpose: Reports on cardiac problems with oral proton pump inhibitors have caused extensive safety reviews by the U.S. Food and Drug Administration. We provide additional data on acute cardiac effects of an intravenous application.

Methods: Echocardiography was performed in 18 healthy volunteers after administration of a common high dose regimen of pantoprazole (80 mg IV bolus followed by 8 mg/h for 1h) or placebo. Design: Randomized, double-blind, placebo-controlled crossover trial.

Results: EF [%, means+/-S.E.] in the treatment group (placebo group) was 60.7+/-1.1 (61.2+/-1.7) at baseline, and 62.6+/-1.1 (62.1+/-1.9), 64.7+/-1.6 (63.5+/-1.3), 62.6+/-1.6 (61.0+/-1.6) and 63.0+/-1.4 (61.8+/-1.5) at 7.5, 15, 30 and 60 min after bolus application, respectively (p = n.s.). Similarly, no significant changes were found for cardiac output, cardiac index, blood pressure, and heart rate. In contrast, gastric pH that was used as a treatment control was significantly increased 60 min after application of pantoprazole as compared to baseline and to placebo.

Conclusions: Pantoprazole for injection is safe in healthy subjects with respect to cardiac contractile function. However, in view of recent reports of negative inotropy of the drug further studies in heart failure patients are required.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 or < 40 years
* No signs of overt heart failure
* Echocardiographic ejection fraction >= 55%
* Body Mass Index 20 - 25 kg/m²
* Excellent sonographic conditions
* Non-smoker
* Informed consent

Exclusion Criteria:

* History of cardiac disease
* History of other relevant pre-existing illness
* Pathologic findings in clinical examinations
* Pathologic echocardiographic findings
* Pathologic ECG findings
* Pathologic laboratory findings
* Pregnancy and lactation
* No or insufficient contraception
* Intolerance of pantoprazole
* Alcohol or drug abuse

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-05; Primary Completion 2006-01 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Echocardiographic ejection fraction | 60 min

SECONDARY OUTCOMES:
Cardiac index | 60 min

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Hasenfuss, Prof. Dr., Principal Investigator — Herzzentrum Goettingen
Locations (1):
- Dept. of Cardiology and Pneumology; Herzzentrum Goettingen, Göttingen, Germany

REFERENCES:
- [Result] Schillinger W, Hornes N, Teucher N, Sossalla S, Sehrt D, Jung K, Hunlich M, Unsold B, Geiling B, Ramadori G, Hilgers R, Schworer H, Hasenfuss G. Recent in vitro findings of negative inotropy of pantoprazole did not translate into clinically relevant effects on left ventricular function in healthy volunteers. Clin Res Cardiol. 2009 Jun;98(6):391-9. doi: 10.1007/s00392-009-0012-6. Epub 2009 Mar 20. PMID 19301059